CLINICAL TRIAL: NCT00194922
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study of the Tolerance and Efficacy of the Probiotic E. Coli Strain M17 on Symptoms and Quality of Life in Individuals With Irritable Bowel Syndrome (IBS)
Brief Title: Study to Determine the Effectiveness of the Probiotic E. Coli Strain M17 in Treating Irritable Bowel Syndrome (IBS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: BioBalance Corporation (Industry)
Responsible Party: Robert Hoerr, The BioBalance Corporation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BB-03-02003
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2008-04-04 (Estimated); Status verified 2008-04

CONDITIONS: Irritable Bowel Syndrome (IBS)
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Placebo Comparator)
  Interventions: Dietary Supplement: E. Coli Strain M17 Probiotic

INTERVENTIONS:
Dietary Supplement: E. Coli Strain M17 Probiotic — 30 ml PO BID for 12 weeks
  Other Names: ProBactrix

SUMMARY:
The purpose of this study is to determine the tolerance and efficacy of the probiotic E. Coli Strain M17 on symptoms and Quality of Life in Individuals with Irritable Bowel Syndrome (IBS).

DETAILED DESCRIPTION:
IBS is characterized by abdominal discomfort and altered bowel function, without identifiable structural or biochemical abnormalities. Current management approaches are not satisfactory for many individuals, who continue to have intermittent constipation or diarrhea, associated with abdominal discomfort.

Probiotics, or "friendly bacteria", is the name given to a new category of products that show promise for managing the symptoms of IBS. In the intestine they are believed to compete with other bacteria, to product substances that interfere with other bacteria, and to improve the function of the mucous lining and immune function of the gastrointestinal tract. A common source of probiotics is in cultured dairy products,m such as yogurt or cheese. E. coli Strain M17 is not regulated vy the Food and Drug Administration. It is considered to be a health food supplement.

E. coli strain M17 was identified in Russia more than 70 years ago. It became widely used in countries of the former Soviet Union for a variety of gastrointestinal problems, including IBS, inflammatory bowel disease (ulcerative colitis or Crohn's disease), and diarrhea, including infants and children. It continues to be produced and marketed under government control in the Russian Federation. E. coli strain M17 was brought to Israel in the early 1990's by two Russian scientists. It was developed for human use and animal feed and approved for use by the Israeli health authorities. A special liquid formulation was developed and sold as a nutritional supplement in pharmacies in Israel until 2002 when the product was acquired by a U.S. company, the BioBalance Corporation, for the purpose of introducing it outside Israel as a medical food and nutritional supplement in the U.S. and other countries.

The purpose of this research study is to compare the tolerability and effectiveness of E. coli strain M17 to placebo in the treatment of Irritable Bowel Syndrome (IBS).

ELIGIBILITY:
Inclusion Criteria:

* Age =18 or =80, males and females.
* Diagnosed with IBS by Rome II criteria , also called "bloating"
* Normal colonic anatomy in the past 5 years as evidenced by a colonoscopy, flex sigmoidoscopy, Barium enema, Sonography, or other exam deemed acceptable by the study physician
* Normal thyroid function tests (or compensated on thyroid replacement) and negative antibody screening test for celiac disease.
* Normal blood chemistries and CBC for age, sex measured within 6 months of starting study.

Exclusion Criteria:

* Pregnant, breast-feeding, or not using approved methods of contraception (if of childbearing potential)
* Unstable medical disorder or other GI disorder (per discretion of screening physician), especially Crohn's disease, history of carcinomas of the bowel, malabsorption syndrome, intolerance to certain food types (such as lactose), functional diarrhea, and functional constipation
* Patient has undergone MAJOR abdominal surgery in the past (note: an appendectomy, for example, is not included in this definition.
* Patient has had E. coli strain M17 administered in the past six months
* History of major psychiatric disorder or substance abuse within the previous 2 years, including psychiatric illnesses requiring medication that may cause doubt in the validity of the signed Informed Consent form --
* Existing illness or medical condition that will prevent the patient from participating in the study (such as severe heart disease, insulin dependent diabetes, hyperactive thyroid gland, HIV positive, anemia, etc.)
* Participation in another clinical study during the past four weeks.
* Candidate will not be available for the next 18 weeks (2 weeks run-in, 12 weeks study, 4 weeks follow-up)
* Recent abnormal values in any routine lab tests prior to beginning the trial product, with values deviating from normal in either direction by a factor of 2.5, unless follow up test has been shown to be normal. Elevated liver function tests: aspartate aminotransferase or alanine aminotransferase >2.5 times upper limit of normal. Elevated renal function test: serum creatinine > 152.4 mmol/L (or appropriate upper cutoff per lab. Abnormal CBC indicating anemia by age and sex standards. Abnormal urinalysis (evidence of infection or albumin). Hyperthyroidism or hypothyroidism: T4 or TSH greater than or less than normal range. If previously diagnosed, disease must be managed and stable.
* Positive antibody test for celiac disease.
* Non-skin malignancy in previous 5 years
* Any use of an investigational drug within 30 days of screening period
* Any use of a probiotic supplement within 30 days of the screening period (with the exception of standard food yogurt products)
* Any use of antibiotics within 42 days of the screening period (however, candidate may wait to initiate screening exam until 42 days have lapsed since antibiotic course was completed)
* Current use of any drugs or treatments which the study physician believes has caused gastrointestinal symptoms that may be confused with or add to the symptoms of IBS.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2004-08; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Relief of pain and discomfort for at least 2 weeks per month over a 12 week period | at the completion of the study

SECONDARY OUTCOMES:
Changes in stool consistency, stool frequency, and bloating | At the completion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Christine Frissora, MD, Principal Investigator — Weill Medical College of Cornell University; Mark B Pochapin, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Cornell Weill Medical College, New York, New York, United States